CLINICAL TRIAL: NCT07265973
Title: PREPARE: Perioperative REhabilitation Around Vaginal Prolapse RepAir Surgery for Recovery Enhancement
Acronym: PREPARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Sarah Jeney, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-258
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Physical Functioning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Perioperative Care (No Intervention): This arm consists of control subjects who are not assigned to an intervention
- Home Exercise Program (Experimental): This arm consists of subjects who are assigned to perform the home exercise intervention
  Interventions: Other: Pelvic floor Home Exercise Program, this intervention is comprised of specific exercises that are easy to complete at home

INTERVENTIONS:
Other: Pelvic floor Home Exercise Program, this intervention is comprised of specific exercises that are easy to complete at home — Many exercise regimens focus on strengthening your pelvic floor. The intervention for this study is a novel pelvic floor physical therapy program that focuses on relaxing, stretching, and protecting the pelvic floor.
  Arms: Home Exercise Program

SUMMARY:
Pelvic organ prolapse is a common problem faced by millions of patients in the United States, leading to an estimated 200,000 surgeries per year. The majority of patients in the US undergoing vaginal suspension between the ages of 60-79. Deconditioning and decreased functional status after surgery can be more pronounced in elderly populations. It is important to explore ways to improve postoperative functioning for this vulnerable population.

This research study is about how good your physical functioning is after surgery. The physical functioning we are studying consist of normal daily activities, such as walking up and down stairs. This study is for patients with pelvic organ prolapse who are getting vaginal surgery to correct the prolapse.

By doing this study, we hope to learn more about ways to improve physical functioning after vaginal prolapse repair surgery. Patients will be chosen at random to participate in or not to participate in a home daily exercise program for 6 weeks. We have participants who do not participate in the home exercise program so that we can compare their physical functioning to the participants who do exercise at home. By doing this comparison, we can find out if the home exercise program helps postoperative physical functioning.

If you are in the home exercise group, a possible benefit is to have better physical functioning after surgery. If you are not assigned to the exercise group, the benefit is being a part of a study that could potentially help other women and yourself in the future to have better physical functioning after surgery. Patients will be enrolled in teh study only if they are undergoing specific surgeries at the University of New Mexico to correct their pelvic organ prolapse.

DETAILED DESCRIPTION:
The objective of this study is to compare postsurgical physical functioning after transvaginal native tissue prolapse repair between patients undergoing normal perioperative care and patients utilizing a standardized perioperative pelvic floor home exercise program. This objective will be accomplished by randomizing women undergoing sacrospinous ligament suspension, uterosacral ligament suspension, or the Manchester procedure to standard perioperative care or standard perioperative care accompanied by a home exercise program using a 1:1 randomization ratio.

The central hypothesis is that the use of a perioperative exercise program will improve patients' postoperative physical functioning. The resulting positive impact that could come from this study is a standardized method to improve physical functioning and possibly improve deconditioning for patients undergoing transvaginal prolapse repair.

Studies previously mentioned involving PFPT have a high level of heterogeneity of exercises, and the exercises are individualized. One commonality between many studies utilizing PFPT programs is a large strengthening component. This strengthening consists of contractions of the pelvic floor muscles with home exercises often involving daily sets of pelvic floor muscle contractions. Strengthening exercises consisting of daily contractions were not utilized in this exercise program as data does not support a significant positive impact of these exercises. In cooperation with UNM pelvic floor Physical Therapists we developed a novel home PFPT exercise program focused on relaxing, stretching, and protecting the pelvic floor.

Participants will be assigned to either a home exercise group or a standard care group 1-2 months prior to their surgical date. This assignment will be random using a 1:1 ratio. The intervention group will be assigned daily home exercises, these daily exercises are to be started 2 weeks prior to surgery and continue 4 weeks after surgery. An exercise video and written instructions of all that is in the video will be provided in order for the home exercise group to have guidance on how to perform the exercises correctly. The second group, the control/standard care group, will not be provided with exercises and that group is to do their normal daily activities before and after surgery. The standard care group will be provided exercises 6 weeks after surgery, once their participation in the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are ≥ 18 years of age
* English or Spanish speaking
* Stage 2, 3 or 4 uterovaginal or vaginal vault prolapse.
* Patient scheduled to undergo transvaginal sacrospinous ligament suspension, uterosacral ligament suspension, or Manchester procedure at The University of New Mexico Hospital.

Exclusion Criteria:

* Inability to speak English or Spanish
* Currently enrolled in Pelvic floor physical therapy
* Inability to perform the home exercises
* Dementia
* Inability to fill out questionnaires
* Inability to access video via internet
* Undergoing concomitant surgeries that involve: InterStim, bladder hydrodistension/fulguration, pelvic floor Botox, mesh excision/complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
Postoperative physical functioning | Physical functioning will be assessed at baseline when patint is enrolled. Physical functioning will also be assessed postoperatively at 1, 2, and 6 weeks after surgery.
  Postoperative physical functioning will be assessed using a questionnaire. The specific questionnaire is the Patient Reported Outcomes Measurement Information Systems (PROMIS) Physical Function Short Form 20a.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jeney, MD, Principal Investigator
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No